CLINICAL TRIAL: NCT03924830
Title: Influence of Surface Sealants on the Quality of Posterior Restorations With Bulk Fill Composites
Acronym: SEALBULK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFFBULKSEAL2018
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: dentin bonding agents; tooth sensitivity; composite resin restoration
MeSH Terms: conditions — Dentin Sensitivity | interventions — Dietary Fiber; BisCover; PermaSeal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bulk without Surface Sealant (Active Comparator): 53 teeth will receive restorations using Bulk fill restoration without surface sealant
  Interventions: Procedure: Bulk without surface sealant
- Bulk with Biscover (Experimental): 53 teeth will receive restorations using Bulk fill restoration with Biscover surface sealant
  Interventions: Procedure: Bulk with Biscover
- Bulk with Permaseal (Experimental): 53 teeth will receive restorations using Bulk fill restoration with Permaseal surface sealant
  Interventions: Procedure: Bulk with Permaseal

INTERVENTIONS:
Procedure: Bulk without surface sealant — Adhese SE self-etch adhesive system will be applied according to the manufacturer's instructions in 53 teeth.Then, the Tetric N-Ceram Bulk fill composite will be used in increments of no more than 4 mm, using the bulk restoration technique, and each increment will be photoactivated for 40 seconds.
  Arms: Bulk without Surface Sealant
Procedure: Bulk with Biscover — Adhese SE self-etch adhesive system will be applied according to the manufacturer's instructions in 53 teeth.Then, the Tetric N-Ceram Bulk fill composite will be used in increments of no more than 4 mm, using the bulk restoration technique, and each increment will be photoactivated for 40 seconds. After the restoration is completed, biscover surface sealant will be applied according to the manufacturer's instructions.
  Arms: Bulk with Biscover
Procedure: Bulk with Permaseal — Adhese SE self-etch adhesive system will be applied according to the manufacturer's instructions in 53 teeth.Then, the Tetric N-Ceram Bulk fill composite will be used in increments of no more than 4 mm, using the bulk restoration technique, and each increment will be photoactivated for 40 seconds. After the restoration is completed, Permaseal surface sealant will be applied according to the manufacturer's instructions.
  Arms: Bulk with Permaseal

SUMMARY:
Treatment clinical trial, randomized, controled, parallel, double-blinded, with three groups, that aims to evaluate if there is some advantage in applying surface sealants (Biscover, Bisco, USA or Permaseal, Ultradent, USA) associated with a Bulk Fill Composite (Tetric N-Ceram Bulk Fill, Ivoclar Vivadent,Liechtenstein). Volunteers will be selected and recruited,following inclusion criteria and pre-established exclusion. All volunteers will be informed and sign a term of clarification and consent. 53 enrolled patients will receive 159 Class I or Class II dental restorations, made in three different ways, one from each experimental group (no sealant, or one of the evaluated surface sealants). Occlusal or Proximo-occlusal lesions will receive the selected treatments separated by groups. Group Bulk without surface sealant (BNS), Group Bulk and Biscover (BSB), and Group Bulk and Permaseal (BSP). Immediate post-operative tooth sensitivity will be evaluated after one week. Restorations will be evaluated every 6 months for pain assessment, shape, fractures, staining or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

DETAILED DESCRIPTION:
This is a Treatment clinical trial, randomized, controlled, parallel, double-blinded, with three groups, that aims to evaluate if there is some advantage in applying surface sealants (Biscover, Bisco, USA or Permaseal, Ultradent, USA) associated with a Bulk Fill Composite (Tetric N-Ceram Bulk Fill, Ivoclar Vivadent, Liechtenstein). Volunteers will be selected and recruited, following inclusion criteria and pre-established exclusion. All volunteers will be informed and sign a term of clarification and consent. All 53 enrolled patients will receive 159 Class I or Class II dental restorations, made in three different ways, one from each experimental group, using the same self-etching adhesive system, under the restorations that will use the same bulk fill composite. All patients must have at only 20 teeth in function, must have at only 3 carious lesion in occlusal or proximo-occlusal face in posterior teeth or old restorations in the same faces, with problems, that need to be changed. Those lesions must be more than 2 mm deep, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility. Firstly, the patient will be anesthetized locally with 3% Mepivacaine solution, followed by prophylaxis with pumice powder and water. All cavities will be washed and dried after these procedures for optimal selection of color, using a color scale. Then, the rubber dam isolation of the teeth to be restored will be held. Occlusal or Proximo-occlusal lesions will receive the restorative procedurs in 3 different protocols separated by groups. Group Bulk without surface sealant (BNS): the adhesive system will be used in 53 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, and photoactivated during 10 seconds with Light Emission Diode (LED) light. Then, the Tetric N-Ceram Bulk fill composite will be used in increments of 4 mm, using the bulk restoration technique, and photoactivated for 40 seconds; Group Bulk and Biscover (BSB): adhesive and restorative procedures will be performed as described in group BNS in 53 teeth. After the restorations are concluded, Biscover surface sealant will be applied according to the manufacturer's instructions; Group Bulk and Permaseal (BSP): adhesive and restorative procedures will be performed as described in group BNS in 53 teeth. After the restorations are concluded, Permaseal surface sealant will be applied according to the manufacturer's instructions. Immediate post-operative tooth sensitivity will be evaluated after one week. Restorations will be evaluated every 6 months for pain assessment, shape, fractures, staining or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have at only 20 teeth in function, must have at only 3 carious occlusal or proximo-occlusal lesions, or old restorations that need to be changed, in different teeth. Those lesions must be more than 2 mm deep, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility.

Exclusion Criteria:

* Volunteers with periodontal disease; with gingival bleeding; use of anti-inflammatory drugs in the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Restoration Loss | Five years
  It will be evaluated the increase in the number of losses of dental restorations in the period of five years, verified by periodic visual clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of remaining restorations in the different groups.

SECONDARY OUTCOMES:
Marginal Pigmentation | Five years
  It will be evaluated the increase in the number of dental restorations with marginal pigmentation in the period of five years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.
Post-Operative Hypersensitivity | Five years
  It will be evaluated the increase in the number of dental restorations with dentin hypersensitivity in the period of five years, verified by periodic clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with dentin hypersensitivity in the different groups.
Secondary Caries | Five years
  It will be evaluated the increase in the number of dental restorations with secondary caries in the period of five years, verified by periodic radiographic examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with secondary caries in the different groups.

CONTACTS AND LOCATIONS:
Overall Officials: MARCOS O BARCELEIRO, DDS, PHD, Study Director — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense - School of Dentistry, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbas G, Fleming GJ, Harrington E, Shortall AC, Burke FJ. Cuspal movement and microleakage in premolar teeth restored with a packable composite cured in bulk or in increments. J Dent. 2003 Aug;31(6):437-44. doi: 10.1016/s0300-5712(02)00121-5. PMID 12878027
- [Background] Moorthy A, Hogg CH, Dowling AH, Grufferty BF, Benetti AR, Fleming GJ. Cuspal deflection and microleakage in premolar teeth restored with bulk-fill flowable resin-based composite base materials. J Dent. 2012 Jun;40(6):500-5. doi: 10.1016/j.jdent.2012.02.015. Epub 2012 Mar 3. PMID 22390980
- [Background] Roggendorf MJ, Kramer N, Appelt A, Naumann M, Frankenberger R. Marginal quality of flowable 4-mm base vs. conventionally layered resin composite. J Dent. 2011 Oct;39(10):643-7. doi: 10.1016/j.jdent.2011.07.004. Epub 2011 Jul 27. PMID 21801799
- [Background] van Dijken JW, Pallesen U. Randomized 3-year clinical evaluation of Class I and II posterior resin restorations placed with a bulk-fill resin composite and a one-step self-etching adhesive. J Adhes Dent. 2015 Feb;17(1):81-8. doi: 10.3290/j.jad.a33502. PMID 25625133
- [Background] Bayraktar Y, Ercan E, Hamidi MM, Colak H. One-year clinical evaluation of different types of bulk-fill composites. J Investig Clin Dent. 2017 May;8(2). doi: 10.1111/jicd.12210. Epub 2016 Jan 22. PMID 26800647
- [Background] Costa T, Rezende M, Sakamoto A, Bittencourt B, Dalzochio P, Loguercio AD, Reis A. Influence of Adhesive Type and Placement Technique on Postoperative Sensitivity in Posterior Composite Restorations. Oper Dent. 2017 Mar/Apr;42(2):143-154. doi: 10.2341/16-010-C. Epub 2016 Nov 28. PMID 27892839
- [Derived] Calazans FS, Ferreira TMJ, Naupari-Villasante R, Mendonca RP, Ornellas G, Albuquerque EG, Tardem C, de Miranda MS, Barceleiro MO, Loguercio AD. Influence of surface sealants on the quality of posterior restorations with bulk-fill composites: A 4-year randomized clinical trial. Dent Mater. 2024 Mar;40(3):466-476. doi: 10.1016/j.dental.2023.12.011. Epub 2023 Dec 22. PMID 38142146